CLINICAL TRIAL: NCT07072130
Title: The Effect of Using Two Different Skin Cleansing Cotton Swabs on the Skin Condition of Term Newborns During Diaper Care for Meconium Removal
Brief Title: Skin Condition of Term Newborns During Diaper Care for Meconium Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2025-02/77
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Infant ALL; Skin
Keywords: skin care; diaper care; skin condition assessment; meconium; infant; newborn
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (wet cotton) (Other): The newborns whose meconium-stained diapers were cleaned with wet cotton comprised the control group.
  Interventions: Other: Control group (wet cotton)
- Experimental group (baby oil-impregnated cotton) (Experimental): The newborns whose meconium-stained diapers were cleaned with baby oil-impregnated cotton comprised the experimental group
  Interventions: Other: Experimental group (baby oil-impregnated cotton)

INTERVENTIONS:
Other: Control group (wet cotton) — The diaper area of the newborns in the control group was cleaned using only cottons moistened with boiled and warmed water. In the preparation stage, the cottons were placed in disposable containers and boiled and warmed water was poured over them to moisten the entire surface of the cottons. Excess water was removed by gently squeezing the cottons. After cleaning, the application was completed by drying the gland area with dry cotton.
  Arms: Control group (wet cotton)
Other: Experimental group (baby oil-impregnated cotton) — Diaper area cleaning of newborns in the experimental group was performed only with cottons impregnated with baby oil. In the preparation of these cottons, a sufficient amount of baby oil was added to the cottons placed in disposable containers and the entire surface of the cottons was allowed to absorb the oil. Excess oil was removed by gently squeezing the cottons. After the cleaning process was completed, the diaper area was dried with dry cotton wool and the process was terminated.
  Arms: Experimental group (baby oil-impregnated cotton)

SUMMARY:
The aim of this study was to determine the effect of two different skin cleansing cotton wipes on skin condition during meconium removal diaper care in term newborns.

The following hypotheses were tested: (a) There is no difference between the effect of using wet cotton and baby oil-impregnated skin cleansing cotton on skin condition during meconium removal diaper care in term newborns. (b) There is a difference between the effect of using wet cotton and baby oil-impregnated skin cleansing cotton on skin condition during meconium removal diaper care in term newborns.

DETAILED DESCRIPTION:
Newborns pass a substance called meconium in the first 24-48 hours through feces. Meconium is a sticky substance consisting of epithelial cells containing green, brown and dark colored mucus. Although meconium can be cleaned with soft tissue wipes that do not contain alcohol and odor or cotton soaked with water, it is difficult to clean because of its adhesive structure. Diaper care practices, wiping, rubbing procedures and materials used during care are important parameters that may threaten skin integrity and should be taken into consideration. In the literature, skin disorders in the diaper area are among the most common skin problems encountered by newborns in the first year. The skin of newborns is different from that of adults. The function of the epidermis is not yet complete and studies have reported that it continues to complete the maturation process in the first year of life.

However, the gland area in infants has higher hydration and pH levels than other areas. The change in skin pH affects the ionization level of molecules and topical absorption. Friction and prolonged exposure of this area to feces further increase the skin pH and potentiate the action of skin irritating fecal enzymes. Therefore, it is important to keep the diaper area clean at all times and maintain adequate hydration.

It is an important necessity to develop a special method for easier removal of meconium formed in the first days of life without damaging the skin integrity. In this study, skin condition score was evaluated by using wet cotton and baby oil-impregnated skin cleansing cotton during diaper care for meconium removal.

ELIGIBILITY:
Inclusion Criteria:

* Newborns 38 gestational weeks and older
* Healthy newborns
* Newborns who defecate their first meconium

Exclusion Criteria:

* Newborns with abnormal skin condition
* Newborns with gastrointestinal tract disease
* Newborns with parental history of skin disease
* Newborns with developmental delay
* Newborns with meconium defecation before the first skin assessment

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in score of skin condition | 1 hour after birth; immediately after the first meconium diaper care; 3 hours and 6 hours after the first meconium diaper care.The change in these time period will be measured.
  Skin condition was measured using a validated and reliable skin condition score. The scale consists of three items and each item includes an evaluation criterion. These are dryness, erythema and disruption/peeling of skin integrity, respectively. Each item of the three-point Likert scale is scored from 1 to 3. The lowest score that can be obtained from the scale is 3 and the highest score is 9; a high total score indicates that the skin condition of the newborn is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assoc. Prof., Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusari A, Han AM, Virgen CA, Matiz C, Rasmussen M, Friedlander SF, Eichenfield DZ. Evidence-based skin care in preterm infants. Pediatr Dermatol. 2019 Jan;36(1):16-23. doi: 10.1111/pde.13725. Epub 2018 Dec 12. PMID 30548578
- [Background] Lund CH, Osborne JW. Validity and reliability of the neonatal skin condition score. J Obstet Gynecol Neonatal Nurs. 2004 May-Jun;33(3):320-7. doi: 10.1177/0884217504265174. PMID 15180195
- [Background] Lavender T, Furber C, Campbell M, Victor S, Roberts I, Bedwell C, Cork MJ. Effect on skin hydration of using baby wipes to clean the napkin area of newborn babies: assessor-blinded randomised controlled equivalence trial. BMC Pediatr. 2012 Jun 1;12:59. doi: 10.1186/1471-2431-12-59. PMID 22656391
- [Background] Brandon DH, Hatch D, Barnes A, Vance AJ, Harney J, Voigtman B, Younge N. Impact of diaper change frequency on preterm infants' vital sign stability and skin health: A RCT. Early Hum Dev. 2022 Jan;164:105510. doi: 10.1016/j.earlhumdev.2021.105510. Epub 2021 Nov 20. PMID 34896732
- [Background] Gustin J, Bohman L, Ogle J, Fadayel G, Mitchell MC, Narendran V, Visscher MO, Carr AN. Improving newborn skin health: Effects of diaper care regimens on skin pH and erythema. Pediatr Dermatol. 2021 Jul;38(4):768-774. doi: 10.1111/pde.14602. Epub 2021 May 31. PMID 34060142